CLINICAL TRIAL: NCT02560051
Title: Phase 2 Study of Androgen Deprivation Therapy (ADT) Plus Chemotherapy as Initial Treatment for Local Failures or Advanced Prostate Cancer
Brief Title: Hormone Therapy Plus Chemotherapy as Initial Treatment for Local Failures or Advanced Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual; resource re-allocation
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert J Amato, Director and Professor, Department of Internal Medicine, Division of Oncology, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU-13-101; HSC-MS-14-0949 (Other: UTHSC-H Committee for Protection of Human Subjects)
Record Dates: First submitted 2015-09-17; First posted 2015-09-25 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Advanced; Local Failures
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Doxorubicin; Ketoconazole; Docetaxel; Estramustine; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Definitive local therapy (Active Comparator): 3 cycles of chemotherapy (doxorubicin, ketoconazole, docetaxel and estramustine) + 12 months ADT (degarelix)
  Interventions: Drug: Doxorubicin; Drug: Ketoconazole; Drug: Docetaxel; Drug: Estramustine; Drug: Degarelix
- Nodal only/Low-volume bone (Active Comparator): 4 cycles of chemotherapy (doxorubicin, ketoconazole, docetaxel and estramustine) + 18 months ADT (degarelix)
  Interventions: Drug: Doxorubicin; Drug: Ketoconazole; Drug: Docetaxel; Drug: Estramustine; Drug: Degarelix
- High volume/no prior tx (Active Comparator): 5 cycles of chemotherapy (doxorubicin, ketoconazole, docetaxel and estramustine) + 24 months ADT (degarelix)
  Interventions: Drug: Doxorubicin; Drug: Ketoconazole; Drug: Docetaxel; Drug: Estramustine; Drug: Degarelix

INTERVENTIONS:
Drug: Doxorubicin — In weeks 1, 3, and 5 of each 8-week cycle, participants will receive doxorubicin (20 mg/m2 as a 24-hour intravenous infusion on day 1 of each applicable week)
  Other Names: Adriamycin; Rubex
Drug: Ketoconazole — In weeks 1, 3, and 5 of each 8-week cycle, participants will receive ketoconazole (400 mg orally 3 times daily for 7 days)
  Other Names: Nizoral
Drug: Docetaxel — In weeks 2, 4, and 6 of each 8-week cycle, participants will receive docetaxel (35 mg/m2 intravenously on day 1 of each applicable week)
  Other Names: Taxotere; Docecad
Drug: Estramustine — In weeks 2, 4, and 6 of each 8-week cycle, participants will receive estramustine (280 mg orally 3 times daily for 7 days)
  Other Names: Emcyt
Drug: Degarelix — The starting dose (240 mg given as two injections of 120 mg each) is followed by maintenance doses of 80 mg administered as a single injection every 28 days
  Other Names: Firmagon

SUMMARY:
This study is for men who have prostate cancer and have failed local therapy or are not a candidate for prostatectomy or radiation therapy. The purpose of this research study is to assess the safety and benefit of androgen deprivation therapy (ADT, blocks hormones) plus chemotherapy. Degarelix is the hormone blocking drug that will be used. Doxorubicin, Ketoconazole, Docetaxel and Estramustine are the chemotherapy drugs that will be used. The drugs used in this study are approved by the Food and Drug Administration (FDA).

Participants will be treated with ADT plus chemotherapy for three, four, or five 8-week cycles (12, 18, or 24 months). The number of cycles of chemotherapy they receive and the number of months they receive ADT will be based on their disease. The current standard treatment is ADT and chemotherapy. What differs in this research study is the cycling and combination of chemotherapy drugs chosen. The drugs chosen for this study have fewer side effects and are believed to provide maximum benefit.

DETAILED DESCRIPTION:
As a working hypothesis, investigators suspect that the transformation from an androgen-dependent to an androgen-independent phenotype is mediated by expansion of an androgen-independent clone already present at the time of ADT that continues to grow while androgen-sensitive clones are being suppressed. It is thus desirable to bring treatment to bear on the androgen-independent component while the corresponding tumor burden remains minimal and prolong the time to hormone resistance. Investigators view the androgen-independent component as analogous to "microscopic residual" or "micro-metastatic" disease, for which adjuvant chemotherapy has been shown to be effective in other contexts, even when the same drugs had little or no impact on survival in the setting of more advanced disease.

By treating all components of the tumor initially, investigators anticipate that the emergence of androgen-independent growth will be delayed, ultimately prolonging patient survival. Additionally, instead of treating patients empirically with an identical regimen, as in investigator's previous work, these patient subsets were designed to ensure a level of treatment appropriate to their individual disease, thus potentially lessening the burden of treatment (such as the long-term adverse effects of ADT). Investigators have chosen 3, 4, or 5 cycles of chemotherapy to be administered on the basis of tumor burden, a treatment selection method long established in germ cell tumors and used by this PI. Sub-analyses of previous data have raised the concern that treating patients with varying levels of disease the same way does not produce optimal results. Therefore, investigators seek to improve outcomes by tailoring treatment to tumor burden. In this study, patients with less tumor burden will receive 3 cycles of chemotherapy and 12 months of ADT, those with moderate tumor burden will receive 4 cycles and 18 months of treatment, and those with the greatest tumor burden will receive 5 cycles and 24 months of treatment. Additionally, this regimen of administering treatment sequentially, including a 2-week break, reduces toxicity.

ELIGIBILITY:
Inclusion criteria:

* Pathologic proof of adenocarcinoma of the prostate.
* Patients must belong to one of the following subsets:
* Prior local therapy
* Patients with Prostate Specific Antigen (PSA) recurrence following prostatectomy or radiation therapy who have no radiographic involvement. PSA doubling time ≤6 months.
* Nodal involvement only.
* Low volume bone disease: ≤3 metastases.
* Nodal involvement with associated bone involvement.
* High volume bone-visceral disease: Patients with >3 metastatic bone sites or visceral metastases.
* No prior definitive local therapy
* Tumors felt to be unresectable, not candidates for radiation therapy, and PSA elevated with biopsy-proven disease.
* Metastatic disease at presentation.
* Patients may have started ADT within 3 months of study entry.
* No previous cytotoxic therapy is allowed, including systemic irradiation with strontium-89, samarium, or radium-223.
* Previous definitive radiotherapy to one metastatic site is acceptable, provided that unirradiated sites remain. At least 8 weeks must have elapsed since radiation therapy to the pelvis. Patients having limited irradiation of a metastatic site are eligible 4 weeks following radiation.
* Patients may have had previous exposure to ADT if it was given for ≤6 months to "downstage" the primary and provided that such therapy was completed at least 12 months prior to entry into this study with a return of serum testosterone to ≥200 ng/dL.
* Patients must be free of serious comorbidity and have a life expectancy of ≥3 years.
* Patients must have adequate physiologic reserves as evidenced by:
* Eastern Cooperative Oncology Group (ECOG) status of ≤2.
* Patients must have adequate bone marrow function: Platelets ≥100,000 cells/mm3, Hemoglobin ≥9.0 g/dL, and Absolute Neutrophil Count (ANC) ≥1,500 cells/mm3.
* Patients must have adequate renal function: creatinine ≤2 × upper limit of normal (ULN).
* Patients must have adequate liver function: Aspartate aminotransferase (AST) / Alanine transaminase (ALT) ≤2.5 × ULN; alkaline phosphatase <2.5 × ULN, unless bone metastasis is present in the absence of liver metastasis; and bilirubin < ULN or 1.5 mg/dl.
* No evidence of active ischemia on electrocardiogram (ECG) and documentation of ejection fraction (EF) ≥50%.

Exclusion criteria:

* Patients must not have a second malignancy unless there is confidence of previous curative therapy.
* Patients with a recent history of transient ischemic attack (TIA) (within 6 months), who are requiring regular antianginal therapy, or who are having claudication sufficient to limit activity are not eligible. Patients with a previous history of deep venous thrombosis or pulmonary embolism (within 12 months) are not eligible
* Patients must not have a serious intercurrent medical or psychiatric illness, including serious active infection.
* Patients must not have sensory neuropathy > grade 1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Started | 6 | 8 | 5
Completed | 3 | 4 | 4
Not Completed | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx | Total
Number analyzed (Participants) | 6 | 8 | 5 | 19
Age, Continuous [Median (Full Range); unit: years] | 66.5 [54 to 73] | 71 [65 to 80] | 60 [55 to 84] | 68 [54 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 5 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 1 | 0 | 2
  Caucasian | 5 | 6 | 4 | 15
  Hispanic | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 5 | 19
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status scale measures level of functioning. The scale ranges from 0 to 5, with 0 indicating the highest level of functioning and 5 the lowest.
  Participants
    0 | 6 | 5 | 2 | 13
    1 | 0 | 3 | 3 | 6
    2 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by Number Who Progressed
Description: Progression defined as increase in Prostate Specific Antigen (PSA) >0.3 ng/mL over 2 measurements or larger/new lesion
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
Participants | 0 | 0 | 2

2. Secondary Outcome: Efficacy as Measured by Number of Participants With Pathology/Biopsy Positive for Disease
Time Frame: about 10 months after treatment initiation
Population: Fewer were analyzed than the number that started or completed the study because not all participants were biopsied following treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 3 | 3

3. Secondary Outcome: Efficacy as Measured by PSA Level
Description: Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are reported as nanograms of PSA per milliliter (ng/mL) of blood.
Time Frame: baseline
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
ng/mL | 5.7 [0.1 to 27.7] | 15.8 [0.8 to 46.6] | 90.7 [17.5 to 2191]

4. Secondary Outcome: Efficacy as Measured by PSA Level
Description: as for outcome 3
Time Frame: Cycle 1 Day 1, which is the day of treatment initiation
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
ng/mL | 5.7 [0.01 to 27.7] | 9.7 [0.8 to 46.6] | 90.7 [17.5 to 90.7]

5. Secondary Outcome: Efficacy as Measured by PSA Level
Description: as for outcome 3
Time Frame: Cycle 2 Day 1, which is about 8 weeks after treatment initiation
Population: Fewer were analyzed than the number that started study because not all participants completed the full number of cycles of treatment assigned. For some participants treatment was prematurely discontinued at different points through the course of treatment because of adverse events, progression, and participant withdrawal from study.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 7 | 5
ng/mL | 0.01 [0.01 to 0.3] | 0.3 [0.1 to 0.6] | 3.8 [0.6 to 68.1]

6. Secondary Outcome: Efficacy as Measured by PSA Level
Description: as for outcome 3
Time Frame: Cycle 3 Day 1, which is about 16 weeks after treatment initiation
Population: as for outcome 5
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 5 | 6 | 4
ng/mL | 0.01 [0.01 to 0.3] | 0.1 [0.1 to 0.8] | 0.9 [0.3 to 7.0]

7. Secondary Outcome: Efficacy as Measured by PSA Level
Description: as for outcome 3
Time Frame: Cycle 4 Day 1, which is about 24 weeks after treatment initiation
Population: This time point is after 4 cycles of chemotherapy so no one in group "definitive local therapy" were analyzed. For the other groups fewer were analyzed than the number that started study because for some participants treatment was prematurely stopped at different points in treatment because of adverse events, progression, and withdrawal from study.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 0 | 5 | 4
ng/mL |  | 0.01 [0.01 to 0.1] | 0.55 [0.2 to 4.1]

8. Secondary Outcome: Efficacy as Measured by PSA Level
Description: as for outcome 3
Time Frame: Cycle 5 Day 1, which is about about 32 weeks after treatment initiation
Population: This time point is after 5 cycles of chemo so so no participants in the groups that had only 3/4 cycles were included. For the other group fewer were analyzed than the number that started study because for some treatment was prematurely stopped at different points in treatment because of adverse events, progression, and withdrawal from study.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 0 | 0 | 3
ng/mL |  |  | 0.5 [0.1 to 2.6]

9. Secondary Outcome: Efficacy as Measured by PSA Level
Description: Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are reported as nanograms of PSA per milliliter (ng/mL) of blood.
  The time point is the end of treatment, which is about about 8 weeks after the start of the last cycle. For the arm completing 3 cycles, the time point is 24 weeks after treatment initiation. For the arm completing 4 cycles, the time point is 32 weeks after treatment initiation. For the arm completing 5 cycles, the time point is 40 weeks after treatment initiation.
Time Frame: end of treatment, which is about about 8 weeks after the start of the last cycle
Population: Fewer were analyzed than the number that started study because some participants were taken off study at different points in treatment or follow-up because of adverse events, progression, and withdrawal from study.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 7 | 5
ng/mL | 0.01 [0.01 to 0.2] | 0.01 [0.01 to 0.2] | 1.4 [0.1 to 34.4]

10. Secondary Outcome: Efficacy as Measured by Number Who PSA Progressed
Description: PSA progression defined as increase in Prostate Specific Antigen (PSA) >0.3 ng/mL over 2 measurements
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
Participants | 0 | 0 | 1

11. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: The Functional Assessment of Cancer Therapy-Prostate (FACT-P) scale is a tool used for assessing the health-related quality of life (QoL) in men with prostate cancer. It consists of 27 core items which assess patient function in four domains (Physical, Social/Family, Emotional, and Functional well-being), and it is further supplemented by 12 site specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce a global QoL score, with a range of scores of 0 to 156. Higher scores represent better QoL.
Time Frame: post cycle 1, which is about 8 weeks after treatment initiation
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
units on a scale | 97 [62 to 135] | 99 [87 to 123] | 105 [58 to 115]

12. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: as for outcome 11
Time Frame: post cycle 2, which is about 16 weeks after treatment initiation
Population: as for outcome 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 5 | 6 | 5
units on a scale | 94 [62 to 114] | 97 [85 to 124] | 102 [58 to 121]

13. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: as for outcome 11
Time Frame: post cycle 3, which is about 24 weeks after treatment initiation
Population: Fewer were analyzed than the number that started study because some participants were taken off study at different points throughout the study because of adverse events, progression, and participant withdrawal from study. Additionally, some participants did not wish to complete the FACT-P questionnaire.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 1 | 5 | 4
units on a scale | 79 [79 to 79] | 94 [89 to 123] | 114 [101 to 121]

14. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: as for outcome 11
Time Frame: post cycle 4, which is about 32 weeks after treatment initiation
Population: This is after 4 cycles of chemo so no one in group "definitive local therapy" were analyzed. For the other groups fewer were analyzed than the number that started study because for some participants treatment or follow-up was prematurely stopped at different points because of adverse events, progression, and withdrawal from study.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 0 | 3 | 4
units on a scale |  | 96 [93 to 126] | 113 [99 to 121]

15. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: as for outcome 11
Time Frame: post cycle 5, which is about about 40 weeks after treatment initiation
Population: as for outcome 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 0 | 0 | 4
units on a scale |  |  | 107 [89 to 117]

16. Secondary Outcome: Quality of Life Measure by FACT-P Scale
Description: The Functional Assessment of Cancer Therapy-Prostate (FACT-P) scale is a tool used for assessing the health-related quality of life (QoL) in men with prostate cancer. It consists of 27 core items which assess patient function in four domains (Physical, Social/Family, Emotional, and Functional well-being), and it is further supplemented by 12 site specific items to assess for prostate-related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce a global QoL score, with a range of scores of 0 to 156. Higher scores represent better QoL.
  The time point is about 12 weeks after completion of the last cycle. For the arm completing 3 cycles, the time point is 36 weeks after treatment initiation. For the arm completing 4 cycles, the time point is 44 weeks after treatment initiation. For the arm completing 5 cycles, the time point is 52 weeks after treatment initiation.
Time Frame: about 12 weeks after completion of the last cycle
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 3 | 4 | 2
units on a scale | 94 [83 to 115] | 118 [92 to 142] | 99 [93 to 105]

17. Secondary Outcome: Safety of Drug Regimen as Measured by Number of Adverse Events
Time Frame: as for outcome 1
Measure: Number; unit: adverse event
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
Number analyzed (Participants) | 6 | 8 | 5
adverse event | 115 | 270 | 166

ADVERSE EVENTS:
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 10 months.
Arm/Group | Definitive Local Therapy | Nodal Only/Low-volume Bone | High Volume/no Prior tx
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/8 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Definitive Local Therapy (N=6) | Nodal Only/Low-volume Bone (N=8) | High Volume/no Prior tx (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (3) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders, Pulmonary inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Definitive Local Therapy (N=6) | Nodal Only/Low-volume Bone (N=8) | High Volume/no Prior tx (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders, Inverted T-wave on EKG (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders, Red eyes (Eye disorders) | 0 (0) | 1 (4) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (6) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 7 (12) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 4 (6) | 2 (2)
Gastroesophageal Reflux (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (3)
Gastrointestinal Disorders, Loose stools (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 2 (3) | 3 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (9) | 6 (10) | 3 (4)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 5 (11) | 3 (4)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 5 (7) | 7 (11) | 3 (8)
Fever (General disorders) | 1 (1) | 2 (4) | 2 (3)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions, Foot irritation/infection (General disorders) | 0 (0) | 1 (3) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection Site Reaction (General disorders) | 1 (1) | 2 (2) | 2 (3)
Irritability (General disorders) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
Infections and Infestations, Thrush (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (5) | 2 (3) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0) | 3 (3)
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 3 (4) | 2 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 5 (11) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders, Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 4 (9) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 1 (2)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (3)
Dysguesia (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (4) | 3 (5)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Nervous system Disorders, Disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (2)
Psychiatric disorder, Emotional (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Renal and urinary disorders, Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders, Penile irritation (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders, Nasal discharge (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders, Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures, Soreness at site (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2) | 1 (1)
Cardiac disorders, Atherosclerotic Ulcer in Posterior Arch of Aorta (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders, Decreased vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders, Discharge from eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders, tongue changes (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorders, Abdominal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders, Motion sickness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders, Body aches/pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
General disorders, Facial/Lip irritation (General disorders) | 2 (2) | 0 (0) | 0 (0)
General disorders, Mental Fogginess/Forgetfulness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders, Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal and urinary disorders, Urinary burning (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders, Dry nostrils (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders, Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders, Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02560051/Prot_SAP_000.pdf